CLINICAL TRIAL: NCT00003494
Title: Phase II Study of Antineoplastons A10 and AS2-1 In Patients With Bronchial Alveolar Carcinoma of the Lung
Brief Title: Antineoplaston Therapy in Treating Patients With Recurrent or Stage IV Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066533; BC-LA-5 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Bronchial Alveolar; Tumor
Keywords: Bronchial Alveolar Cancer Recurrent; Bronchial Alveolar Cancer Stage IV
MeSH Terms: conditions — Neoplasms | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with Recurrent or Stage IV Lung Cancer will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)ANP

SUMMARY:
Current therapies for Recurrent or Stage IV Lung Cancer provide very limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Recurrent or Stage IV Lung Cancer.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Recurrent or Stage IV Lung Cancer.

DETAILED DESCRIPTION:
Recurrent or Stage IV Lung Cancer patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Recurrent or Stage IV Lung Cancer, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Recurrent or Stage IV Lung Cancer.
* To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or stage IV bronchoalveolar cell lung cancer unlikely to have a curative response to existing standard regimens
* Measurable disease by MRI or CT scan

  * At least 2 cm in diameter

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No renal insufficiency
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No severe heart disease
* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease (e.g., chronic obstructive pulmonary disease)

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections
* No other concurrent serious disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Recovered from prior surgery

Other:

* No prior antineoplaston therapy
* Prior cytodifferentiating agent allowed

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 1996-03-26 (Actual); Primary Completion 2002-05-26 (Actual); Study Completion 2002-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com